CLINICAL TRIAL: NCT04964882
Title: Effect of the Peak Inspiratory Pressure and Facial Mask Holding Techniques on the Gastric Insufflation During Positive Pressure Ventilation With Facemask in Obese Adults
Brief Title: Gastric Insufflation During Positive Pressure Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 31-2021
Record Dates: First submitted 2021-03-31; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Gastric Insufflation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- C-E Mask ventilation under PIP 10 cmH2O (Experimental): Two-handed C-E technique is performed during face mask ventilation using a mechanical ventilator with a peak inspiratory pressure of 10 cmH2O.
  Interventions: Diagnostic Test: ultrasound examination of air insufflation in the upper esophageal region and stomach
- C-E Mask ventilation under PIP 15 cmH2O (Experimental): Two-handed C-E technique is performed during face mask ventilation using a mechanical ventilator with a peak inspiratory pressure of 15 cmH2O.
  Interventions: Diagnostic Test: ultrasound examination of air insufflation in the upper esophageal region and stomach
- C-E Mask ventilation under PIP 20 cmH2O (Experimental): Two-handed C-E technique is performed during face mask ventilation using a mechanical ventilator with a peak inspiratory pressure of 20 cmH2O.
  Interventions: Diagnostic Test: ultrasound examination of air insufflation in the upper esophageal region and stomach
- V-E Mask ventilation under PIP 10 cmH2O (Experimental): Two-handed V-E technique is performed during face mask ventilation using a mechanical ventilator with a peak inspiratory pressure of 10 cmH2O.
  Interventions: Diagnostic Test: ultrasound examination of air insufflation in the upper esophageal region and stomach
- V-E Mask ventilation under PIP 15 cmH2O (Experimental): Two-handed V-E technique is performed during face mask ventilation using a mechanical ventilator with a peak inspiratory pressure of 15 cmH2O.
  Interventions: Diagnostic Test: ultrasound examination of air insufflation in the upper esophageal region and stomach
- V-E Mask ventilation under PIP 20 cmH2O (Experimental): Two-handed V-E technique is performed during face mask ventilation using a mechanical ventilator with a peak inspiratory pressure of 20 cmH2O.
  Interventions: Diagnostic Test: ultrasound examination of air insufflation in the upper esophageal region and stomach

INTERVENTIONS:
Diagnostic Test: ultrasound examination of air insufflation in the upper esophageal region and stomach — Presence of air insufflation is assessed using ultrasound in the upper esophageal region and stomach during face mask ventilation

SUMMARY:
Effect of peak inspiratory pressure on the gastric insufflation is evaluated using ultrasonography during face mask ventilation in obese adults. Effect of facial mask holding techniques on the gastric insufflation is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with body mass index ≥ 30 kg/m2 who are scheduled for general anesthesia

Exclusion Criteria:

* Risk of delayed gastric emptying or gastroesophageal reflux (gastroesophageal reflux disease, achalasia, history of stomach surgery, gastrointestinal obstruction, uncontrolled DM)
* Pregnancy
* Known or predicted difficult airway

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-07-20 (Estimated); Primary Completion 2022-03-05 (Estimated); Study Completion 2022-03-05 (Estimated)

PRIMARY OUTCOMES:
Presence of gastric insufflation in the epigastric region | During anesthesia induction
  Under ultrasound, air signal is assessed in the epigastric region

SECONDARY OUTCOMES:
Cross-sectional area of the antral cross-sectional area | During anesthesia induction
  During ultrasound examination, anterior-posterior diameter and cranio-caudal diameter of the antrum are measured. Cross-sectional area of the gastric antrum is calculated as follows; (AP × CC × π)/4 (AP=antero-posterior diameter and CC=cranio-caudal diameter).
Presence of gastric insufflation in the upper esophageal region | During anesthesia induction
  Under ultrasound, air signal is assessed in the upper esophageal region.
Expiratory tidal volume | During anesthesia induction
  Expiratory tidal volumes displayed on the monitor of the anesthesia machine are recorded.